CLINICAL TRIAL: NCT00261092
Title: Phase II Multicenter, Open Label Study of Oxaliplatin Combined With Gemcitabine(GEMOX) in Advanced and Metastatic Pancreatic Cancer
Brief Title: GEMOX: Oxaliplatin in Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM_L_0126
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin

SUMMARY:
Primary objective:

* To evaluate overall response rate (based on RECIST criterion)

Secondary objective:

* To evaluate time to progression, clinical benefit, quality of life and safety

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the pancreas
* Metastatic or locally advanced, non resectable disease(Non resectable disease will be determined by the investigators with clinical data)
* Uni-dimensionally measurable disease as defined by RECIST (primary or secondary tumors>2cm using conventional CT scan or ≥1cm with spiral CT scan)
* No previous chemo or radiotherapy, but postoperative radiotherapy as a adjuvant therapy for non-target lesion is permitted
* Karnofsky Performance Status (KPS) ≥60
* No known Central Nervous System metastases
* No sensory neuropathy at inclusion
* Biological and hematological evaluation < 2 weeks prior to treatment administration:

  * Neutrophils ≥ 1500/ mm3
  * Platelets ≥ 100,000/mm3
  * Alkaline phosphatases< 5X ULN(upper Limits of Normal) and Bilirubin < 1.5X ULN
  * SGOT,SGPT <2.5 X ULN if no liver metastasis
  * SGOT,SGPT <5 X ULN if liver metastasis
  * Creatinine < 1.5 X ULN
* Baseline imaging (CT scan or Magnetic Resonance Imaging) <3 weeks before treatment administration
* Men and women who are fertile must use a medically acceptable contraceptive throughout the treatment period and for 3 months following cessation of treatment with oxaliplatin. Subjects must be made aware, before entering this trial of the risk of becoming pregnant or in fathering children

Exclusion Criteria:

* Corticotherapy except for anti-emetic purpose
* Pregnant or breast feeding women (Documentation of a negative pregnancy test must be available for premenopausal women with intact reproductive organs)
* Uncontrolled congestive heart failure or angina pectoris, or hypertension or arrhythmia
* Uncontrolled or persistent hypercalcemia
* History of significant neurologic or psychiatric disorders
* Vater ampulomas and biliary tract adenocarcinomas
* Other -non cured- malignancies

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2005-10

PRIMARY OUTCOMES:
Overall response rate based on RECIST criteria

SECONDARY OUTCOMES:
Time to progression
Overall survival
Clinical benefit
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Won-Sik Lee, MD, Study Director — sanofi-avents
Locations (1):
- Sanofi-Aventis, Seoul, South Korea